CLINICAL TRIAL: NCT04331665
Title: A Single Arm Open-label Clinical Study to Investigate the Efficacy and Safety of Ruxolitinib for the Treatment of COVID-19 Pneumonia
Brief Title: Study of the Efficacy and Safety of Ruxolitinib to Treat COVID-19 Pneumonia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A Phase III RUXCOVID study evaluating ruxolitinib on top of standard of care (SoC) therapy compared to SoC treatment alone in patients with COVID-19 did not meet its primary endpoint. With this news, recruitment was stopped for this study.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-DEPLOY: RUX-COVID; 20-5315 (Other: University Health Network)
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib to prevent COVID-19 pneumonia (Experimental): All participants will receive ruxolitinib at at 10 mg, twice a day, for 14 days, followed by 5 mg, twice a day, for 2 days and 5 mg, once daily, for 1 day.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is an inhibitor of JAK1 and JAK2 (proteins important in cell signalling) approved for the treatment of myelofibrosis, polycythemia vera, and graft-versus-host disease.
  Other Names: JAKAVI

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the drug ruxolitinib in people diagnosed with COVID-19 pneumonia by determining the number of people whose conditions worsen (requiring machines to help with breathing or needing supplemental oxygen) while receiving the drug.

This is a sub-study of the U-DEPLOY study: UHN Umbrella Trial Defining Coordinated Approach to Pandemic Trials of COVID-19 and Data Harmonization to Accelerate Discovery. U-DEPLOY helps to facilitate timely conduct of studies across the University Health Network and other centers.

DETAILED DESCRIPTION:
Multifocal interstitial pneumonia is the most common cause of deterioration in people with COVID-19. This is attributed to a severe reaction where releases too many cytokines (proteins that play an important role in immune responses) which rush into the lungs resulting in lung inflammation and fluid buildup. This can lead to damage to the lungs and leading to breathing problems. Ruxolitinib when given early in the disease, may prevent the overproduction of cytokines which, in turn, may prevent lung damage.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection diagnosed by nasopharyngeal sample
* Need for supplemental oxygen to maintain oxygen saturation > 93%
* 12 years of age or older

Exclusion Criteria:

* Neutrophils < 1 x 10^9/L
* Platelets < 50 x 10^9/L
* Serum total bilirubin >2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST), or alanine aminotransferase (ALT) > 5x ULN
* Creatinine clearance (CrCl) < 15 mL/minute
* Pregnant women
* Known HBV or HIV infection
* Signs and symptoms of Varicella Zoster Virus (VZV) infection
* Patients requiring invasive mechanical ventilation. Patients requiring non-invasive mechanical ventilation (e.g., BiPAP) are eligible.
* Patients who require supplemental oxygen support prior to COVID-19 infection.
* Patients who are on ruxolitinib or similiar drugs.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with COVID-19 pneumonia who become critically ill (defined as requiring mechanical ventilation and/or FiO2 of 60% of more) | 6 months
Number of adverse events | 9 months

SECONDARY OUTCOMES:
All cause mortality rate | 9 months
Average duration of hospital stay | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chan, M.D., Principal Investigator — Princess Margaret Cancer Centre; Vikas Gupta, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kramer A, Prinz C, Fichtner F, Fischer AL, Thieme V, Grundeis F, Spagl M, Seeber C, Piechotta V, Metzendorf MI, Golinski M, Moerer O, Stephani C, Mikolajewska A, Kluge S, Stegemann M, Laudi S, Skoetz N. Janus kinase inhibitors for the treatment of COVID-19. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD015209. doi: 10.1002/14651858.CD015209. PMID 35695334